CLINICAL TRIAL: NCT05074576
Title: The Effect of Mulligan Mobilization Technique Application in Addition to Classical Therapies on Pain and Joint Range of Motion People With Neck Pain
Brief Title: The Effect of Mulligan Mobilization Technique
Acronym: TheEffect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, ozluozge, MSc, PT, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ozluozge
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Orthopedic Disorder of Spine; Manual Therapy; Physical Therapy
Keywords: Mulligan Mobilization; Mechanical Neck Pain
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are blind for allocation and outcomes measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan group (Experimental): In addition to the conventional treatments, Sustained Natural Apophysial Gliding (SNAG) a type of Mulligan mobilization technique is applied.
  Interventions: Other: Mulligan group
- Control group (Other): Electroterapy agents are applied in the contro group
  Interventions: Other: Control group

INTERVENTIONS:
Other: Mulligan group — Ultrasound (8minutes, 1.5 w/cm2, pulsed), conventional transcutaneous electrical nerve stimulation (TENS) (20 minutes, 60-120 Hz frequency) and hot pack application (20 minutes) and interferential current (100 rpm) as electrotherapy agents. In addition to the conventional treatments, Sustained Natural Apophysial Gliding (SNAG) a type of Mulligan mobilization technique is applied. Mobilization is performed by giving 15-20 seconds rest between 3 sets of 4-5 repetations.
  Patients were treated in a sitting position. SNAG technique was applied by the physiotherapist at each on spinal level. Active movement with using passive manual force in the direction of translation or rotation was applied to the cervical vertebrae. At the end range of the joint, overpressure was applied by the patient himself
  Arms: Mulligan group
Other: Control group — Electroterapy agents are applied in the same conditions with Mulligan Group. Active neck, shoulder and thoracic region exercises for correction postural misalignment are performed in both groups. All exercises were done in 3 sets of 10 repetitions. Stretching exercises of upper part of Trapezius, sternocleidomastoideus and pectoral muscles are done with 10 repetitions and for 15-30 seconds.
  Arms: Control group

SUMMARY:
The aim of this study is to investigate the effect of the Mulligan mobilization technique on pain intensity and range of motion individuals with neck pain. The patients were randomized into two groups. Group 1 is the Mulligan Mobilization group and the second group is the control group.

DETAILED DESCRIPTION:
The study is designed as a single-center, parallel-group, randomized controlled clinical trial in Istanbul Medipol university hospital.

The study will be conducted on 40 volunteers with mechanical neck pain. The patients were randomized into two groups. Groups were determined by randomization method with closed box. A random paper was drawn for the participants included in the study.

Inclusion criterias are being between age of 25-65 years, having neck pain for at least 2 weeks, participants that were diagnosed with MNP by a doctor, having no contraindicated condition for manual treatment. Exclusion criterias were surgical indications and/ or surgery history for cervical region, history of trauma to the cervical region and those with systemic disease, participation of physical therapy and rehabilitation program in the last one year, fibromyalgia, presence of cardiac pacemaker, intra-articular steroid injection in neck joint in the last three months.

In the intervention; Mulligan mobilization technique, electroterapy and active range of motion and stretching exercises carried out in Mulligan group while only electrotherapy agents and exercises are applied as a classical treatment to the control group. Goniometer for the range of motion of the neck (ROM), Visual Analogue Scale (VAS), Neck Pain And Disability Scale (NPDS), Short Form Health Survey (SF-36) will be used for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Being between age of 25-65 years,
* having neck pain for at least 2 weeks,
* participants that were diagnosed with MNP by a doctor,
* having no contraindicated condition for manual treatment.

Exclusion Criteria:

* surgical indications and/ or surgery history for cervical region,
* history of trauma to the cervical region and those with systemic disease,
* participation of physical therapy and rehabilitation program in the last one year,
* fibromyalgia,
* presence of cardiac pacemaker,
* intra-articular steroid injection in neck joint in the last three months.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-10-15 (Estimated); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
Range of Motion | 10 minutes
  Universal goniometer is used to measure the joint position and joint range of motion measurements based on Kendall and American Association of Orthopedic Surgeons. The participant is in the sitting position and asked to perform active cervical region flexion, extension, right and left rotation, right and left lateral flexion of the neck movements and performed degrees are recorded.
Pain status | 5 minutes
  Pain intensity is evaluated with visual analog scale (VAS) in two conditions during activity and resting time. This method, which is developed to determine the intensity of pain to indicate by numbers. It begins with the absence of pain (0) on numerical scale and ends the level of unbearable pain
Life quality | 15 minutes
  Quality of life of the participants are evaluated by Short Form 36 (SF-36). It is a self-assessment scale developed by Rond Corporation in 1992. Short Form 36 (SF-36) is a personalized scale that assesses the general health status of the patients with 36 questions, 8 Sub-Items (Physical function, physical role weakness, body pain, general health, vitality, social function, emotional function, mental function). SF-36 scale is scored from 0 to 100 (0 = worst, 100 = best)
Disability status | 10 minutes
  The items assess the severity of pain and the relationship between pain, occupational, social, recreational, emotional factors. It determines the effect of neck pain on disability, functionality and quality of life. Total score is the sum of the points in each item and ranges from 0 to 100. High scores indicate that more affected status

CONTACTS AND LOCATIONS:
Overall Officials: OZGE OZLU, Principal Investigator — Medipol University
Locations (1):
- Ozge Ozlu, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
When I will publish this manuscript in a journal, I would share the results of individual participant data of this study with other researchers.

REFERENCES:
- [Result] Ganesh GS, Mohanty P, Pattnaik M, Mishra C. Effectiveness of mobilization therapy and exercises in mechanical neck pain. Physiother Theory Pract. 2015 Feb;31(2):99-106. doi: 10.3109/09593985.2014.963904. Epub 2014 Sep 29. PMID 25264016
- [Derived] Ozlu O, Sahin M. The effect of mulligan mobilization technique application in addition to conventional physiotherapy on pain and joint range of motion in people with neck pain. J Bodyw Mov Ther. 2024 Jul;39:225-230. doi: 10.1016/j.jbmt.2024.02.009. Epub 2024 Mar 5. PMID 38876630